CLINICAL TRIAL: NCT00943969
Title: Determinants of Oral Morphine Answer Among Obese Patients Before and After Gastric Bypass
Acronym: OBEMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia LLORET LINARES, MCU-PH, Hopital Lariboisière
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CPP 0911965
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: obesity; gastric bypass; morphine; pharmacokinetic; absorption
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- obemo (Other)
  Interventions: Procedure: gastric bypass

INTERVENTIONS:
Procedure: gastric bypass — gastric bypass combines restrictive and malabsorptive procedures

SUMMARY:
The bariatric surgery is widely used to treat obesity. Roux-en-Y gastric bypass is one of the most frequently surgical methods performed and combines restrictive and malabsorptive procedures. Different data suggest that this surgery may modify drug absorption and we think it would be clinically relevant to describe the consequences of gastric bypass on drug systemic exposure in obese patients, since no data on the comparison between the pharmacokinetics (PK) of a drug before and after surgery are available and help to predict the drugs posology.The investigators decided to study the morphine because there is a lack of information about the PK, pharmacodynamics (PD) et pharmacogenetics (PG) of morphine in obese subjects, in contrary with anaesthetic drugs. This is a drug with a narrow therapeutic range frequently prescribed in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years old.
* Patients with morbid obesity (IMC > 40 kg/m²) or severe obesity (IMC=35-40 kg/m²) with co morbidities (sleep apnea syndrome or hypertension or steatosis hepatitis) with a favourable decision of a multidisciplinary team for a gastric bypass.
* Patient agreeing to go 3 times for a one day hospitalisation in the URT of the Lariboisière Hospital for the morphine PK/PD.
* Patient with a previous medical examination.
* Patient giving its well-informed and free consent after information.

Exclusion Criteria:

* diabetes
* concomitant sedative, antidepressive or analgesic treatments or drugs unadvised with morphine
* untreated sleep apnea syndrom, hypoxia (PaO2<70mmHg) or hypercapnia (PaCO2>45mmHg), anaemia <10g/dL, ASAT or ALAT>3N

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
30mg Oral morphine systemic exposure (AUC 0-24) | Before surgery-7-15 days after surgery- 6 months after surgery

SECONDARY OUTCOMES:
Morphine and M6G AUC, clearance, Cmax and Tmax | Before surgery-7-15 days after surgery- 6 months after surgery
fat mass and total body water (assessed by DEXA and BIA) | before surgery and 6 months following surgery
mRNA and protein expression of P-gp , UGT2B7, MRP2 and MRP3 in intestinal biopsies | obtained from the bariatric surgery
genetic polymorphisms known to affect expression and/or activity of enzymes, receptors and transporters involved in morphine PK/PD (UGT2B7, P-gp, OPRM1, COMT) and morphine PK/PD | Before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Célia LLoret Linares, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Unit of Therapeutic Research, Department of Internal Medicine, Lariboisière Hospital, Paris, France